CLINICAL TRIAL: NCT04326465
Title: Fractionated Carbon Dioxide Laser Therapy for Treatment of Peyronie's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ryan Flannigan, MD, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H18-02482
Record Dates: First submitted 2019-08-12; First posted 2020-03-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Peyronies Disease
Keywords: Peyronies Disease; Fractionated Carbon Dioxide Laser
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Intervention Model Description: Efficacy and safety trial for Fractional CO2 Laser Therapy with pre- and post-treatment comparisons (3 laser therapy sessions over 12 weeks in men with Peyronie's Disease).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Fractional CO2 Laser Therapy at 10-15% Laser Density Coverage (Experimental): Study participants with Peyronies Disease will be treated with a Fractional Carbon Dioxide Laser set at a 10-15% laser density. The patient will receive three laser therapy sessions over 12 weeks (one session every four weeks). Following each session, topical triamcinolone will be applied to the treated area.
  Interventions: Device: Fractional Carbon Dioxide Laser Therapy at 10-15% Laser Density Coverage

INTERVENTIONS:
Device: Fractional Carbon Dioxide Laser Therapy at 10-15% Laser Density Coverage — Fractional Carbon Dioxide Laser Therapy is an ablative therapy where abnormal collagen in scarred tissue is destroyed to permit the formation of more organized collagen. Previous studies have demonstrated its efficacy in treating medical conditions (ex. hypertrophic scars) similar to Peyronies Disease. There is evidence that Fractional Carbon Dioxide Laser Therapy has the ability to target and alter the molecular pathways that are similar to the ones that lead to Peyronie's Disease.

SUMMARY:
This is a pilot study that evaluates the use of Fractional Carbon Dioxide Laser Therapy in the treatment of Peyronie's Disease. Study participants will be assigned to receive Fractional Carbon Dioxide Laser Therapy at 10-15% laser density coverage.

DETAILED DESCRIPTION:
Peyronie's Disease is a fibrosing disorder of the penis where scar tissue known as a "plaque" forms along the shaft of the penis. This plaque can lead to penile deformity, erectile dysfunction and pain during intercourse. Furthermore, Peyronie's Disease has been shown to negatively affect the quality of life and cause psychosocial distress. Currently, treatments for Peyronie's Disease are invasive (injections or surgery). This study investigates the use of a non-invasive and extra-dermal Fractional Carbon Dioxide Laser Therapy to treat chronic phase Peyronie's Disease.

Fractional Carbon Dioxide Laser Therapy works by destroying and reducing abnormal collagen (a major component found in Peyronie's Disease plaques) in scarred tissue. Although Fractional Carbon Dioxide Lasers have yet to be used in the field of urology, it has already been used safely and successfully to treat conditions similar to Peyronie's Disease (ie. hypertrophic burn scars).

Study participants enrolled in this study will be required to attend 6 study visits. The first study visit is a 'Screening Visit'. At this visit, a medical history and baseline penile measurements (degree of curvature, stretched length, and circumference deformity at flaccid and erect states) will be collected. Study participants will also be asked to complete the International Index of Erectile Function Questionnaire and Peyronie's Disease Questionnaire.

Following the 'Screening Visit', study participants will be scheduled for three Fractional Carbon Dioxide Laser Therapy sessions. These sessions will be scheduled once every six weeks (totalling 12 weeks from the first therapy session).

Following, the last Fractional Carbon Dioxide Laser Therapy session, there will be three follow-up appointments (Week 18, Week 24, Week 52). At these visits, post-therapy penile measurements, International Index of Erectile Function, and Peyronie's Disease scores will be collected.

Digital photographs may be taken as part of the study's analysis and to track the progress of Fractional CO2 Laser Therapy. You will have the option to deny any digital photography.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males age 18 or older in a stable relationship with a female partner/spouse (for at least 3 months and willing to have vaginal intercourse with that female partner/spouse.
2. Diagnosis of Peyronie's Disease for at least 12 months with evidence of stable disease as determined by the investigator.
3. Penile curvature of 30º-90º in the dorsal, lateral, or dorsal/lateral plane (must have been possible to delineate the single plane of maximal curvature for evaluation).
4. Signed informed Ethics-approved consent agreement; signed authorization form to allow disclosure of protected information.
5. Ability to read, complete, and understand the various rating instruments in English.

Exclusion Criteria:

1. Penile curvature of <30º or >90º.
2. Any conditions affecting the penis such as a chordee in the presence or absence of hypospadias; thrombosis of the dorsal penile artery; infiltration by a benign or malignant mass or an infectious agent; ventral curvature from any cause; presence of an active sexually transmitted disease; known active hepatitis B or C; known immune deficiency disease (including Human Immunodeficiency Virus).
3. Failure to achieve a sufficient erection (after prostaglandin or Trimix administration), in the opinion of the investigator, to accurately measure the penile deformity.
4. Calcified plaque as evident by appropriate radiographic evaluation, i.e. penile ultrasound that would prevent treatment with Fractional Carbon Dioxide Laser.
5. Isolated hourglass deformity of the penis without curvature.
6. Treatment or plans to undergo treatment for Peyronie's Disease, including but not limited to any previous surgery, oral/topical agents within 3 months, intralesional medical therapies within 3 months, extracorporeal shock wave therapy within 6 months, or use of mechanical devices within 2 weeks before the start of the study.
7. Use of or plans to use a mechanical devices to induce a passive erection within 2 weeks before the start of study.
8. Erectile dysfunction that was unresponsive to Phosphodiesterase inhibitors.
9. Received an investigation drug or treatment within 30 days before start of the study.
10. At any time, received Collagenase clostridium histolyticum for the treatment of Peyronie's Disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Measured reduction in penile curvature | Change in penile measurements (Baseline vs. Week 18, 24, & 52).
  Penile measurements will be collected at erect states. Penile measurements will be conducted at the screening visit (Baseline) and at the follow-up study visits (Week 18, 24, & 52).

SECONDARY OUTCOMES:
International Index of Erectile Function Questionnaire | Change in International Index of Erectile Function Questionnaire score (Baseline vs. Week 18, 24, & 52).
  Self-reported 15-item questionnaire that assesses erectile dysfunction. Each item is scored from 0 to 5, yielding a total of 0 to 75.
Peyronie's Disease Questionnaire | Change in Peyronie's Disease Questionnaire score (Baseline vs. Week 18, 24, & 52).
  Self-reported 15-item questionnaire that assesses sexual function in individuals with Peyronie's Disease. Scoring of each item is varied (ie. Q1 scored 0 to 4, Q9 scored 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Flannigan, MD, Principal Investigator — UBC Faculty of Medicine - Department of Urologic Sciences
Locations (1):
- Diamond Health Care Centre, Vancouver, British Columbia, Canada